CLINICAL TRIAL: NCT05060276
Title: A Phase 1B, Dose-Escalation Study of the Safety and Preliminary Efficacy of an Anti-Trop2 Antibody Drug Conjugate (STI-3258) in Patients With Relapsed or Refractory Solid Tumors
Brief Title: Study to Assess an Anti-Trop2 Antibody Drug Conjugate in Relapsed or Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol changed to Phase 2
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2ADC-RRST-101
Record Dates: First submitted 2021-08-20; First posted 2021-09-29 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Relapsed Solid Neoplasm; Refractory Cancer; Solid Tumor, Adult
Keywords: relapsed or refractory solid tumors
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: To determine DLT and MTD, the design uses a 3+3 ascending dose cohort design evaluating up to five dose cohorts including: 8 mg/kg, 12 mg/kg, 16 mg/kg, 20 mg/kg, 24 mg/kg.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-3258 (Experimental): Intravenous infusion to be given with prophylaxis for infusion reactions, evaluating up to five dose cohorts including: 8 mg/kg, 12 mg/kg, 16 mg/kg, 20 mg/kg, and 24 mg/kg.
  Interventions: Biological: STI-3258

INTERVENTIONS:
Biological: STI-3258 — Intravenous infusion of STI-3258 will be given (one infusion every three weeks).
  Other Names: anti-Trop2-SN38 antibody drug conjugate (ADC)

SUMMARY:
This is a phase 1b, open-label, dose-escalation study o STI-3258 administered intravenously in subjects with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose-escalation study o STI-3258 administered intravenously in subjects with relapsed or refractory solid tumors including ovarian, breast, lung, esophageal, gastric, hepatocellular and urothelial cancers.

The study will determine any dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), assessing safety and preliminary efficacy using ascending dose cohorts and a conventional 3+3 study design.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced cancer that is relapsing or refractory to at least one prior treatment and not a candidate for other treatments or is intolerant to established treatments.
* At least one measurable disease per Response Evaluation Criteria in Solid Tumors v. 1.1 (RECIST 1.1).
* Eastern Cooperative Oncology Group Performance Status ≤ 2.
* Must have a life expectancy of ≥ 6 months.
* Must have adequate bone marrow, hepatic and renal function as assessed by specific laboratory tests.
* Must be recovered ≤ Grade 1 from acute toxicities from previous therapies, excluding alopecia and vitiligo.
* Has not had prior treatment within 2 weeks of screening with high dose corticosteroids.
* Be willing and able to comply with the study schedule and all study requirements.
* Willing to follow all contraception guidelines.

Exclusion Criteria:

* Previous treatment with any systemic therapy or investigational drug within 2 weeks of the first dose of study drug.
* Currently participating in any other interventional clinical study.
* Has a diagnosis of other malignancies if the malignancy has required therapy within the last 3 years or is not in complete remission.
* Has presence of bulky disease defined as any mass > 7 cm in greatest dimension will trigger a discussion with the medical monitor.
* Has left ventricular ejection fraction (LVEF) < 40%.
* New York Heart Association (NYHA) Class ≥ 3.
* Has prolonged QTcF interval on an electrocardiogram.
* Has spinal cord compression or clinically active brain metastases.
* Has a history of Sacituzumab govitecan treatment.
* History of anaphylactic reaction to irinotecan or ≥ Grade 3 toxicity to prior irinotecan treatment.
* Has active or prior COVID-19 infection, with symptoms presenting within 4 weeks of the first dose of study drug.
* Has an active bacterial, viral, or fungal infection.
* Is currently pregnant or breast feeding or planning on either during the study.
* Has chronic or moderate chronic obstructive pulmonary disease or other chronic respiratory conditions unless receiving treatment and stable for 3 months prior to screening.
* Has known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C.
* Has any significant medical condition, abnormality, or psychiatric illness that would prevent study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of adverse events (AEs) by type, frequency, severity, and causality
Incidence of treatment-emergent adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of treatment-emergent AEs (TEAEs) by type, frequency, severity, and causality
Incidence of serious adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of serious AEs (SAEs) by type, frequency, severity, and causality
Incidence of Infusion-related adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of Infusion-related AEs (IrAEs) by type, frequency, severity, and causality
Incidence of dose-limiting toxicities (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of dose-limiting toxicities
Determine the MTD | Baseline through study completion at up to approximately 24 months
  Determine the MTD of STI-3258
Determine the RP2D | Baseline through study completion at up to approximately 24 months
  To determine the RP2D of STI-3258

SECONDARY OUTCOMES:
Assess preliminary efficacy of STI-3258 | Baseline through study completion at up to approximately 24 months
  To assess the preliminary efficacy of STI-3258 in the treatment of patients with RRSTs based upon Response evaluation criteria in solid tumors (RECIST).
Assess the area under the curve (AUC) pharmacokinetic profile of STI-3258 | Baseline through study completion at up to approximately 24 months
  To assess the AUC of STI-3258 in plasma as a measure of exposure to the ADC, STI-3258.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.